CLINICAL TRIAL: NCT02313220
Title: A 24-week, Single Centre, Randomized, Parallel-group, Double-blind, Placebo Controlled Phase II Study With an Optional 28-week Open-label Extension to Evaluate the Efficacy on Body Weight of Dapagliflozin 10 mg Once Daily in Combination With Exenatide 2 mg Once Weekly in Obese Non-diabetic Subjects.
Brief Title: Exploratory Study to Investigate the Effect of Dapagliflozin and Exenatide Combined on Body Weight
Acronym: Dapalost
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1690L00016; 2014-003432-39 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Obesity; Dapagliflozin; Exenatide; Combination treatment; Type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin and exenatide (Experimental): Dapagliflozin 10 mg film-coated tablet once daily and exenatide 2 mg once weekly injection combined treatment for 24 weeks
  Interventions: Drug: Dapagliflozin; Drug: Exenatide
- Placebo (Placebo Comparator): Placebo film-coated tablet once daily and placebo once weekly injection combined treatment for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Oral use
  Other Names: Forxiga®
  Arms: Dapagliflozin and exenatide
Drug: Exenatide — Powder and solvent for suspension for injection, prolonged release suspension. Subcutaneous use.
  Other Names: BYDUERON®; BYETTA®
  Arms: Dapagliflozin and exenatide
Drug: Placebo — Oral and Subcutaneous use.
  Arms: Placebo

SUMMARY:
Obesity is a medical condition which increases the risk of other diseases, such as type 2 diabetes and cardiovascular disease. Obesity-related risk factors for the development of other metabolic diseases include unstable glucose levels and high blood pressure. Dapagliflozin and exenatide are both approved worldwide for treatment of patients with Type 2 Diabetes. Dapagliflozin works by lowering glucose levels by inhibiting the renal reabsorption of glucose and thereby promoting its urinary excretion and energy loss and thereby reduction in body fat. Exenatide exhibits many of the same glucose-lowering actions of that of a naturally occurring hormone and leads to weight loss mainly via reduced energy intake, most likely via a central effect on appetite regulation. The purpose of this exploratory study is to investigate if a combination treatment with dapagliflozin and exenatide have a synergistic effect on weight loss in non-diabetic obese subjects. Subjects will be treated for 24 weeks with either active combination treatment or placebo (non-active treatment). Neither study personnel nor subjects will know what treatment is given. All subjects completing the 24-week double-blind study and who are willing and eligible will be offered to enter a 28-week open-label extension study. All subjects entering the extension study will receive unblinded active study treatment for an additional 28 weeks. Thus the total treatment period for subjects entering the extension study will be 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent prior to any study specific procedures.
2. Female and/or male aged 18 to 70 years with body mass index (BMI) (measured as body weight (kg)/(height (m))2) 30 to 45 kg/m2.
3. Female subjects must meet all of the following criteria:

   1. Not breastfeeding
   2. Negative pregnancy test result (human chorionic gonadotropin, beta subunit [beta hCG]) at Visit 1 (Enrolment) (not applicable to hysterectomized females).
   3. If of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year), must practice and be willing to continue to practice one of the following highly effective birth control methods during the entire duration of the study:

      * Diaphragm or partner use of condom in combination with combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

        * Oral
        * Intravaginal
        * Transdermal
      * Diaphragm or partner use of condom in combination with progestogen-only hormonal contraception associated with inhibition of ovulation:

        * Oral
        * Injectable
        * Implantable
      * Placement of an intrauterine device
      * Placement of an intrauterine hormone-releasing system
      * Bilateral tubal occlusion
      * Vasectomised partner (provided that the partner is the sole sexual partner of the female subject and that the vasectomised partner has received medical assessment of the surgical success)
      * Sexual abstinence (defined as refraining from heterosexual intercourse)
   4. Must practice appropriate birth control as stated above for 10 weeks after the last dose of study medication

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study.
2. Previous enrolment in the present study.
3. Participation in another clinical study with an Investigational Product during the last 3 months prior to Visit 1.
4. History of any clinically significant disease, disorder or condition which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
5. Previously diagnosed diabetes mellitus; or fasting P-glucose ≥7.0 mmol/L at Visit 1 confirmed by one more measurement; or P-glucose ≥11.1 mmol/L at 120 min of the oral glucose tolerance test (OGTT) at Visit 1 confirmed by one more measurement. Note: Subjects with a fasting P-glucose of ≥7.0 mmol/L at Visit 1 or ≥11.1 mmol/L at 120 min of the OGTT at Visit 1 may be offered an extra visit before Visit 2 for a second fasting P-glucose measurement. If P-glucose is still ≥7.0 mmol/L at the second measurement, the subject will be excluded.
6. Any clinically significant abnormalities in physical examination or clinical chemistry results as judged by the investigator. The following specific exclusion criteria apply to the selected Clinical Chemistry results:

   1. Creatinine clearance <60 mL/min (estimated with Cockcroft-Gault formula).
   2. Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN.
   3. Total bilirubin (TB) >2.0 mg/dL (34.2 µmol/L).
7. Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody Immunoglobulin M (IgM), Hepatitis B surface antigen and Hepatitis C virus antibody.
8. Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
9. Acute Coronary Syndrome (ACS) within 2 months prior to Visit 1. Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment. Acute Stroke or transient ischemic attack (TIA) within two months prior to Visit 1. Less than two months post coronary artery revascularization.
10. History of gastroparesis or pancreatitis
11. History of malignancy within the last 5 years, excluding successful treatment of basal or squamous cell skin cancer.
12. Body weight loss greater than 5% within 3 months prior to Visit 1.
13. Treatment with any drug known to affect body weight within the last month, e.g. systemic glucocorticoids, antipsychotics or orlistat.
14. Multiple Endocrine Neoplasia syndrome type 2.
15. Personal or family history of medullary thyroid carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | From randomization to 24 weeks
  To assess the efficacy of dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination compared to placebo on body weight after 24 weeks of treatment in obese subjects

SECONDARY OUTCOMES:
Body weight (%) | From randomization to 24 weeks
  To assess the efficacy of dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination compared to placebo on body weight after 24 weeks of treatment in obese subjects

OTHER OUTCOMES:
Proportion of subjects with at least 10% reduction in weight and proportion of subjects with at least 5% reduction in weight. | From randomization to 24 weeks
  To assess the proportion of subjects responding to treatment with dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination when compared to placebo, with respect to change in body weight
Changes in body fat (%), liver fat (%), liver volume (l), total liver fat (l), visceral adipose tissue (l), subcutaneous adipose tissue (l), total adipose tissue (l) and total lean tissue (l). | From randomization to 24 weeks
  To assess the efficacy of dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination compared to placebo on total body fat mass, total lean body mass, percentage liver fat, visceral fat mass and subcutaneous fat mass.
3 h oral glucose tolerance test, frequently sampled for insulin sensitivity and secretion indices. Changes in glucose, glucagon, glycerol, free fatty acids, insulin and C-peptide. | From enrolment to 24 weeks
  To assess the efficacy of dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination compared to placebo on glucose tolerance, insulin secretion, insulin sensitivity and lipolysis regulation.
Changes in total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides, diastolic blood pressure, systolic blood pressure, pulse, waist circumference and waist-hip ratio. | From enrolment to 24 weeks
  To assess the efficacy of dapagliflozin 10 mg once daily and exenatide 2 mg once weekly in combination compared to placebo on blood lipid profile, blood pressure and other anthropometric measurements.
Obesity-related genotypes and pharmacogenetics. | From enrolment to 24 weeks
  To collect and store DNA for future exploratory research of genes/genetic variation that is related to obesity or to treatment response to dapagliflozin in combination with exenatide.
Adverse events /serious adverse events, vital signs and collection of clinical chemistry/haematology parameters. | From enrolment to 24 weeks
  To evaluate the safety and tolerability of dapagliflozin 10 mg once daily and once weekly 2 mg exenatide in combination in obese non-diabetic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eriksson, Prof., MD, Principal Investigator — Uppsala University
Locations (1):
- Dept of Medical Sciences, Clinical Diabetes and Metabolism, Uppsala University and Section for Diabetes and Endocrinology at the Uppsala University Hospital, Uppsala, Sweden